CLINICAL TRIAL: NCT04017572
Title: Optimized vs. Standard Automated Peritoneal Dialysis Regimens (OptiStAR): A Randomized Controlled Trial
Brief Title: Optimized vs. Standard Automated Peritoneal Dialysis Regimens Study
Acronym: OptiStAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Universidad de Córdoba (Other); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PCT171447
Record Dates: First submitted 2019-07-04; First posted 2019-07-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: End Stage Kidney Disease; Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: dialysis; peritoneal dialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment (Active Comparator): APD-treatment with a net volume of 12 L 1.36 % anhydrous glucose peritoneal dialysis solution during 540 minutes.
  Interventions: Procedure: Automated peritoneal dialysis (APD)
- Optimized treatment (Active Comparator): APD-treatment with a net volume of 14 L 2.27 % anhydrous glucose peritoneal dialysis solution during 280 minutes followed by a net volume of 10 L 0.1 % glucose dialysis fluid during 200 minutes.
  Interventions: Procedure: Automated peritoneal dialysis (APD)

INTERVENTIONS:
Procedure: Automated peritoneal dialysis (APD) — Automated peritoneal dialysis (APD) using the Baxter HomeChoice Pro Cycler.

SUMMARY:
This clinical study is designed to evaluate the theoretical prediction of a lower glucose absorption in optimized automated peritoneal dialysis regimes. Patients will receive both a standard 6 x 2L 1.36% glucose regime or an optimized 7 x 2 L 2.27% glucose + 5 x 2 L 0.1% glucose regime in a crossover fashion.

DETAILED DESCRIPTION:
Automated peritoneal dialysis (APD) is a rapidly growing, home-based kidney replacement therapy promoting patient autonomy, and is associated with lower societal costs compared to hemodialysis. However, in light of the growing number of diabetic patients on PD, the unwanted glucose absorption during APD is problematic. Recent results (Öberg CM, Rippe B, 2017, see references), using a theoretical model of APD, indicate that large reductions in glucose absorption are possible by using specialized so-called optimized bi-modal treatment regimes having "UF cycles" using a higher glucose concentration (e.g. 2.27% glucose) and "Clearance cycles" using a low glucose concentration (e.g. 0.1% glucose).

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years;
* duration of PD (automated peritoneal dialysis (APD) or continuous ambulatory peritoneal dialysis (CAPD)) >4 weeks

Exclusion Criteria:

* severe heart failure (New York Heart Association Functional Classification; NYHA III or IV);
* pregnancy;
* catheter malfunction or
* peritonitis within 3 months prior to the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Glucose absorption | Through study completion, up to 1 year
  Amount of glucose absorbed across the peritoneal membrane during the treatment

SECONDARY OUTCOMES:
Ultrafiltration | Through study completion, up to 1 year
  Amount of water transported from the circulation to the peritoneal cavity during the treatment
Creatinine clearance | Through study completion, up to 1 year
  Amount of creatinine transported from the circulation to the peritoneal cavity during the treatment
Urea clearance | Through study completion, up to 1 year
  Amount of urea transported from the circulation to the peritoneal cavity during the treatment
Sodium removal | Through study completion, up to 1 year
  Amount of sodium transported from the circulation to the peritoneal cavity during the treatment
Incidence of complications | Up to 14 days post-intervention
  Complications that are or can be suspected to be related to the study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Carl M Öberg, M.D., Ph.D., Principal Investigator — Lund University
Locations (1):
- Hospital Privado Centro Médico de Córdoba, Córdoba, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oberg CM, Rippe B. Optimizing Automated Peritoneal Dialysis Using an Extended 3-Pore Model. Kidney Int Rep. 2017 Apr 27;2(5):943-951. doi: 10.1016/j.ekir.2017.04.010. eCollection 2017 Sep. PMID 29270500
- [Derived] Bergling K, de Arteaga J, Ledesma F, Oberg CM. Optimized vs. Standard Automated Peritoneal Dialysis Regimens (OptiStAR): study protocol for a randomized controlled crossover trial. Pilot Feasibility Stud. 2020 Jun 10;6:81. doi: 10.1186/s40814-020-00620-2. eCollection 2020. PMID 32528722